CLINICAL TRIAL: NCT04975581
Title: Rotator Cuff Tears Repair With or Without Dermal Patch Augmentation
Acronym: CUFFPATCH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDGE ID 139197
Record Dates: First submitted 2021-05-06; First posted 2021-07-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotator cuff repair Surgery with Augmentative patch (Experimental): Open rotator cuff repair Surgery with additional application of augmentative human allograft patch
  Interventions: Biological: Allograft Patch
- Rotator cuff repair surgery (Active Comparator): Open Rotator cuff repair surgery
  Interventions: Biological: Allograft Patch

INTERVENTIONS:
Biological: Allograft Patch — Rotator Cuff repair with Allograft Patch (Graftjacket Now)

SUMMARY:
The Investigators are planning to conduct a Pilot study of 40 patients of Pragmatic randomised controlled trial comparing rotator cuff tendons repair (small tendons around the shoulder ) with or without augmentative patch. It includes patients between age groups 50 to 75 years with large (≥ 3cm and < 5 cm ) rotator cuff tear that can be fully repaired using open or mini open repair with or without an augmentation with a human dermal matrix allograft (processed skin graft from a human donor ). The main aim is to examine whether the addition of the patch helps to reduce the rate of re-tear of the rotator cuff tendons at one year following surgery. Patients are randomized to receive either a repair with addition of an augmentative patch or a repair without a patch and have an identical follow-up after surgery. Patients are followed up in outpatient at 6 weeks , 3 months and 12 months after randomization and receive an Magnetic Resonant Imaging (MRI) scan 12 months after surgery. The primary outcome measure is to assess the Re-tear rate of rotator cuff at 12 months after surgery. The secondary outcome measure is to assess functional scores of the shoulder at 12 months . The tertiary outcome measures are to check the cost effectiveness of each procedure.

DETAILED DESCRIPTION:
The Investigators are planning to conduct a Pilot study of 40 patients of Pragmatic randomised controlled trial comparing rotator cuff tendons repair (small tendons around the shoulder ) with or without augmentative patch. It includes patients between age groups 50 to 75 years with large (≥ 3cm and < 5 cm ) rotator cuff tear that can be fully repaired using open or mini open repair with or without an augmentation with a human dermal matrix allograft (processed skin graft from a human donor ). The main aim is to examine whether the addition of the patch helps to reduce the rate of re-tear of the rotator cuff tendons at one year following surgery. Patients are randomized to receive either a repair with addition of an augmentative patch or a repair without a patch and have an identical follow-up after surgery. Patients are followed up in outpatient at 6 weeks , 3 months and 12 months after randomization and receive an Magnetic Resonant Imaging (MRI) scan 12 months after surgery. The primary outcome measure is to assess the Re-tear rate of rotator cuff at 12 months after surgery. The secondary outcome measure is to assess functional scores of the shoulder at 12 months . The tertiary outcome measures are to check the cost effectiveness of each procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged at least 50 years to 75 years.
2. Degenerative cuff tear.
3. Large Full thickness rotator cuff tear (≥ 3cm and < 5 cm ) that is fully repairable.
4. Tears diagnosed using MRI scan.
5. Ability to consent.
6. Agreement to use of human dermal matrix allograft as augmentative patch

Exclusion Criteria:

1. Previous surgery on the affected shoulder.
2. Osteoarthritic changes.
3. Unable to have MRI Scans.
4. Significant neck pathology.
5. Cognitive problems or language issue.
6. Systemic arthritis
7. Significant dual pathology in the involved shoulder
8. Acute Traumatic tears (< 6 months since injury).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Retear on MRI scan | 12-18 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsitals of Leicester NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided